CLINICAL TRIAL: NCT07054879
Title: A Prospective Single-center Observational Study: ctDNA-guided Maintenance Therapy for Postoperative Pancreatic Cancer
Brief Title: CtDNA-guided Maintenance Therapy in Pancreatic Cancer
Status: Recruiting | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Du Juan, Chief Physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: PC-Maintenance therapy
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; maintenance therapy; ctDNA; capecitabine maintenance therapy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumor sample and plasma sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experiment Group: Patients received 6 cycles of standard adjuvant chemotherapy (gemcitabine plus capecitabine), followed by capecitabine monotherapy as maintenance treatment based on the patient's clinical condition

SUMMARY:
This study aims to conduct a large-scale prospective clinical trial to evaluate the efficacy and safety of capecitabine monotherapy as maintenance treatment following standard adjuvant chemotherapy (gemcitabine plus capecitabine) in patients with resectable pancreatic cancer, and to analyze whether ctDNA-MRD testing can guide the selection of postoperative maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, male or female
* Histologically or cytologically confirmed primary diagnosis of pancreatic ductal adenocarcinoma (PDAC)
* No evidence of distant metastasis (M0)
* Underwent R0 radical resection within 3 months prior to enrollment
* ECOG performance status of 0-1
* Life expectancy ≥3 months
* Patient or legal guardian is able to understand the study requirements and willing to provide written informed consent

Exclusion Criteria:

* Prior history of radiotherapy, chemotherapy or surgical treatment for pancreatic cancer
* Concurrent severe organ dysfunction or hematologic disorders
* Tumor involvement of celiac axis or superior mesenteric artery, locally advanced disease, or presence of distant metastases
* Poor general condition deemed unable to tolerate chemotherapy
* History of other malignancies within past 5 years (except adequately treated carcinoma in situ of cervix or basal cell carcinoma of skin)
* Any severe or uncontrolled systemic disease that may affect risk/benefit assessment, including but not limited to: uncontrolled hypertension, active hepatitis B or C infection, HIV infection
* Patient or guardian unable to comprehend study objectives and requirements
* Any other condition that in the investigator's judgment would make the patient unsuitable for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pancreatic caner patients with R0 surgery
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
2-year DFS rate | At the timepoint of 2 years after surgery
  the proportion of cancer patients who remain free of disease recurrence or death from any cause within 2 years after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided